CLINICAL TRIAL: NCT00569855
Title: Intravenous Phenoxybenzamine Use in Pediatric Patients Undergoing Open-Heart Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Carole Hamon, University of Arkansas for Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06611
Record Dates: First submitted 2007-12-06; First posted 2007-12-10 (Estimated); Results first posted 2011-03-01 (Estimated); Last update posted 2011-03-01 (Estimated); Status verified 2011-02

CONDITIONS: Open-heart Surgery; Cardiopulmonary Bypass
MeSH Terms: interventions — Phenoxybenzamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Receive phenoxybenzamine in preparation for cardiopulmonary bypass during open-heart surgery
  Interventions: Drug: Phenoxybenzamine

INTERVENTIONS:
Drug: Phenoxybenzamine — 0.125 to 1 mg/kg given i.v. over 15 to 45 minutes in preparation for cardiopulmonary bypass; may be continued at 0.125 mg/kg/day in ICU
  Other Names: Dibenzyline

SUMMARY:
Cardiopulmonary bypass is done with a machine that does the work of the heart and lungs during open-heart surgery. This study is to determine if intravenous (i.v.) phenoxybenzamine is safe. This drug lowers the blood pressure, making it easier for the cardiopulmonary bypass machine to deliver blood and oxygen to all of the organs and tissues.

ELIGIBILITY:
Inclusion Criteria:

* 0-18 years of age
* weight of less than or equal to 20 kilograms

Exclusion Criteria:

* Parental refusal to give informed consent

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 785 (Actual)
Dates: Start 2001-02; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michiaki Imamura, MD, Principal Investigator — Arkansas Childrens Hospital
Locations (1):
- Arkansas Children's Hospital, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The patient population eligible for enrollment included those pediatric patients 20 kilograms or less in weight undergoing open-heart surgery requiring extracorporeal circulation (cardiopulmonary bypass) at Arkansas Children's Hospital, regardless of their gender or ethnic background
Groups:
- Subjects Who Received Study Drug: Subjects less than 20 kgs who received phenoxybenzamine in preparation for cardiopulmonary bypass during open-heart surgery with a dose range between 0.125mg/kg to 0.5mg/kg
Period: Overall Study
Arm/Group | Subjects Who Received Study Drug
Started | 785 (832 subjects enrolled; however, study records only available for analysis from 2004 =446 subjects)
Completed | 785 (785 subjects treated with study drug)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Subjects Who Received Study Drug
Number analyzed (Participants) | 785
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 785
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 390
  Male | 395
Region of Enrollment [Number; unit: participants]
  United States | 785

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Had Significant Hypotension as Defined in the Protocol as Need for Norepinephrine Dose >0.1mcq/kg/Min in the First 72 Hours Postoperatively
Description: Number of subjects who required Norepinephrine >0.1mcq/kg/min
Time Frame: 72 hours postoperatively
Population: No. of subjects consented = 832; 785 subjects received study drug
Measure: Number; unit: participants
Arm/Group | Subjects Who Received Study Drug
Number analyzed (Participants) | 785
participants | 25

ADVERSE EVENTS:
Arm/Group | Subjects Who Received Study Drug
Serious Adverse Events (participants affected / at risk) | 2
Other Adverse Events (participants affected / at risk) | 0/785
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Subjects Who Received Study Drug
Early Death- defined as death within 72 hours of treatment with study drug (Surgical and medical procedures) | 2/785 (2) — AE=early death as defined as death within 72 hours of treatment; cause of death was not analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No